CLINICAL TRIAL: NCT00256399
Title: A Prospective, Open Label, Study to Assess the Efficacy of Alfuzosin 10 mg Tablet Once a Day in Male Subjects Suffering From Benign Prostate Hypertrophy Associated Lower Urinary Tract Symptoms and Erectile Dysfunction
Brief Title: Uroxatral in Men With Benign Prostate Hypertrophy (BPH) and Erectile Dysfunction (ED)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospitals Cleveland Medical Center (Other)
Collaborators: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: L-9835
Record Dates: First submitted 2005-11-18; First posted 2005-11-21 (Estimated); Last update posted 2022-08-15 (Actual); Status verified 2005-11

CONDITIONS: BPH; Erectile Dysfunction
MeSH Terms: conditions — Erectile Dysfunction | interventions — alfuzosin

INTERVENTIONS:
Drug: Alfuzosin 10 mg

SUMMARY:
Uroxatral (alfuzosin) may not only help BPH symptoms but may also improve sexual function in males with BPH and ED.

DETAILED DESCRIPTION:
The study will consist of a 30 day screening/washout phase at the end of which qualified subjects will be assigned to alfuzosin 10 mg tablets once a day. Subjects will be treated for 90 days. The total duration of the study will be 120 days.

ELIGIBILITY:
Inclusion Criteria:

* Males 45-75 years of age
* Confirmed diagnosis of BPH/lower urinary tract symptoms (LUTS) and ED
* Men with steady partner and who agree to attempt sex once a week.

Exclusion Criteria:

* Prostate cancer
* Prostatitis
* Penile disease
* Cardiac co-morbidity
* Pre-existing co-morbid conditions
* History of sensitivity to the drug or similar drugs
* Enrollment in another clinical trial
* Impaired hepatic function
* Impaired renal function
* Mental conditions rendering subject unable to understand the study
* Subjects not likely to comply with protocol

Ages: 45 Years to 75 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2005-11; Primary Completion 2007-05-08 (Actual); Study Completion 2007-05-08 (Actual)

PRIMARY OUTCOMES:
Evaluate the medication on erection maintenance

SECONDARY OUTCOMES:
Assess effect of Uroxatral on BPH and sexual function using questionnaires

CONTACTS AND LOCATIONS:
Overall Officials: Allen D Seftel, MD, Principal Investigator — University Urologists of Cleveland
Locations (1):
- University Hospitals of Cleveland, Cleveland, Ohio, United States